CLINICAL TRIAL: NCT03109834
Title: Choice of Foods, Weight Loss and Metabolic Changes in Overweight Women Willing to Lose Weight With Dietary/Nutritional Therapy Intervention
Brief Title: Effect of Weight Management Programs on Cardiometabolic Risk Profile in Overweight Women
Acronym: FM-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bonn Education Association for Dietetics r.A., Cologne, Germany (Industry)
Collaborators: FomMed HealthCare AG (Unknown)
Responsible Party: Principal Investigator, Christine Metzner, Professor MD, Christine Metzner, Professor MD, Bonn Education Association for Dietetics r.A., Cologne, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFD-01/FM-01
Record Dates: First submitted 2017-03-29; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Overweight and Obesity; Dyslipoproteinemia
Keywords: Weight Management Programs; Weight loss stabilization; Cardiometabolic risk
MeSH Terms: conditions — Overweight; Obesity; Dyslipidemias | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: 2 parallel arms in weight loss phase and weight stabilization phase (1. randomization at baseline I); 2 parallel arms in weight maintanance phase (2. randomization at baseline II)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meal replacement (MR) group (Active Comparator): Energy-restricted modified diet with MR for weight control dietary supplement: MR shakes, soups or bars. Duration: 3-month weight loss phase (phase 1)
  During weight stabilization phase (phase 2) MR counted to food choice option.
  Interventions: Dietary Supplement: Meal replacement (MR)
- Control (C) group (Other): Energy-restricted modified diet without MR for weight control. Duration: 3-month weight loss phase (phase 1)
  During 3-month weight stabilization phase (phase 2) MR counted to food choice option.
  Interventions: Other: Control (C)
- Verum group (Active Comparator): Specific micronutrient composition with omega-3 fatty acids (capsules)
  Duration: 6-month weight maintenance phase (phase 3)
  Interventions: Dietary Supplement: Verum
- Placebo group (Placebo Comparator): Placebo capsules
  Duration: 6-month weight maintenance phase (phase 3)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Meal replacement (MR) — MR-WL group followed an energy-restricted diet with a balanced variety of nutrient-dense food of approximately 1200 kcal/d and was advised to replace two meals, i.e. breakfast and dinner, every day with two MR shakes, soups or bars and to prepare their own lunch during 3-month weight loss phase (phase 1).
  During 3-month weight stabilization phase (phase 2) MR-S group (MR group during weight stabilization phase) were encouraged to consume a self-directed well-balanced variety of nutrient-dense foods without meal intervention. MR counted to food choice option. The MR-S group was instructed to continue the implemented nutrition advice of weight loss phase.
  Duration: 6 months (phase 1 and phase 2: baseline I - 6.month)
  Arms: Meal replacement (MR) group
Other: Control (C) — During 3-month weight loss phase (phase 1) C-WL group followed an energy-restricted diet with a balanced variety of nutrient-dense food of approximately 1200 kcal/d without MR for weight control.
  During 3-month weight stabilization (phase 2) phase C-S group (C group during weight stabilization phase) were encouraged to consume a self-directed well-balanced variety of nutrient-dense foods without meal intervention. MR counted to food choice option. The C-S group was instructed to continue the implemented nutrition advice of weight loss phase.
  Duration: 6 months (phase 1 and phase 2: baseline I - 6.month)
  Arms: Control (C) group
Dietary Supplement: Verum — Verum: Specific micronutrient composition with omega-3 fatty acids (capsules)
  Verum group followed an energy-restricted diet with a balanced variety of nutrient-dense food of approximately 1500 kcal/d and was advised to consume 3 verum-capsules twice a day (with breakfast and dinner) with 200 ml water during 6-month weight loss maintenance phase (phase 3).
  Duration: 6 months (6.month / baseline II - 12.month)
  Arms: Verum group
Other: Placebo — Placebo group followed an energy-restricted diet with a balanced variety of nutrient-dense food of approximately 1500 kcal/d and was advised to consume 3 placebo-capsules twice a day (with breakfast and dinner) with 200 ml water during 6-month weight loss maintenance phase.
  Placebo contains no micronutrients and omega-3 fatty acids.
  Duration: 6 months (6.month / baseline II - 12.month)
  Arms: Placebo group

SUMMARY:
Aim of this prospective randomized study was to evaluate whether a diet with meal replacements can be as effective as a conventional energy-restricted modified diet on weight loss, body composition and cardiometabolic risk profile in overweight women. Moreover, the impact of these two different weight management strategies was observed on cardiometabolic risk profile after a self-directed weight stabilization phase following the weight loss phase. After that, the effect of a specific micronutrient composition with omega-3 fatty acids versus placebo on cardiometabolic risk was observed during a following phase of weight loss maintenance.

DETAILED DESCRIPTION:
Abdominal obesity, atherogenic dyslipidemia and hypertension are essential risk factors for cardiovascular diseases. Several studies showed favorable effects of weight loss in overweight subjects on cardiometabolic risk profile.

The study was divided into a 3-month weight loss phase (phase 1), a subsequent 3-month phase of weight stabilization (phase 2) and a 6-month phase of weight loss maintenance (phase 3).

For a total of 6 months subjects were randomly assigned to the meal replacement (MR) or control (C) group at baseline I.

During weight loss phase both dietary intervention groups followed an energy-restricted diet with a balanced variety of nutrient-dense food of approximately 1200 kcal/d. The MR-WL group (MR group during weight loss phase) was advised to replace two of three meals every day with meal replacements. The C-WL group (C group during weight loss phase) was advised to follow a conventional energy-restricted modified diet with 15-20% of energy intake in the form of protein, 50-55% of energy intake in the form of carbohydrates and 30% of energy intake in the form of fat. All participants attended ten group training sessions for nutrition education.

During weight stabilization phase all women of MR-S and C-S group (MR and C group during weight stabilization phase) were encouraged to consume a self-directed well-balanced variety of nutrient-dense foods without meal intervention. However, the MR-S and C-S group were instructed to continue the implemented nutrition advice of weight loss phase.

At the beginning of weight loss maintenance phase (baseline II) women were randomly assigned to the verum (specific micronutrient composition with omega-3 fatty acids) group or placebo group. Both groups were encouraged to consume a self-directed well-balanced variety of nutrient-dense foods.

All women participated in an exercise program (fitness walking) on 1-2 days per week during all three phases of the study for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI: between 27.0 and 34.9 kg/m²
* One of the following blood lipids: total cholesterol ≥ 200 mg/dL, LDL-cholesterol ≥ 175 mg/dL, HDL-cholesterol ≤ 50 mg/dL, TG 150-400 mg/dL
* women, 18-60 years

Specific Exclusion Criteria:

* lactose or protein intolerance
* hypo- or hyperthyroidism
* pharmacological treatment of diabetes
* intake of vitamins or mineral supplements
* anticoagulants
* cardiac pacemaker
* contraindications to exercise

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2004-03-25 (Actual); Primary Completion 2007-03-28 (Actual); Study Completion 2007-03-28 (Actual)

PRIMARY OUTCOMES:
Weight loss (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Intervention changes in body weight
Total antioxidant capacity (phase 3) | 6-month dietary intervention (from baseline II to 12th month)
  Intervention changes in total antioxidant capacity
Fasting plasma cortisol concentration (phase 3) | 6-month dietary intervention (from baseline II to 12th month)
  Intervention changes in fasting plasma cortisol concentration

SECONDARY OUTCOMES:
Relative body fat (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Intervention changes in relative body fat
Relative body weight (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Intervention changes in relative body weight
Responder (weight loss > 5%) (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Responder rate after 12 weeks
Waist circumference (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Intervention changes in waist circumference
Total antioxidant capacity (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Intervention changes in total antioxidant capacity
Fasting plasma cortisol concentration (phase 1) | 3-month dietary intervention (from baseline I to 3rd month)
  Intervention changes in fasting plasma cortisol concentration
Relative body fat (phase 3) | 6-month dietary intervention (from baseline II to 12th month)
  Intervention changes in relative body fat
Relative body weight (phase 3) | 6-month dietary intervention (from baseline II to 12th month)
  Intervention changes in relative body weight
Responder (weight loss > 5%) | 12 months (from baseline I to 12th month)
  Responder rate after 12 months
Waist circumference (phase 3) | 6-month dietary intervention (from baseline II to 12th month)
  Intervention changes in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Christine Metzner, Professor MD, Principal Investigator — Bonn Education Association for Dietetics r.A., Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Metzner CE, Folberth-Vogele A, Bitterlich N, Lemperle M, Schafer S, Alteheld B, Stehle P, Siener R. Effect of a conventional energy-restricted modified diet with or without meal replacement on weight loss and cardiometabolic risk profile in overweight women. Nutr Metab (Lond). 2011 Sep 22;8(1):64. doi: 10.1186/1743-7075-8-64. PMID 21939523